CLINICAL TRIAL: NCT00681694
Title: Long-Term Outcomes of Alternative Brachytherapy Techniques for Early Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Metro West Medical Center (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: James Talcott, MD, SM, Massachusetts General Hospital
Other Study IDs: 01-264
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Prostate Cancer
Keywords: brachytherapy; radioactive seed implants
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- MRBT: MRI-assisted brachytherapy, the experimental arm
  Interventions: Radiation: brachytherapy
- USBT1: Standard ultrasound-guided brachytherapy performed by group 1 (control arm 1)
  Interventions: Radiation: brachytherapy
- USBT2: Standard ultrasound-guided brachytherapy performed by group 2 (control group 2)
  Interventions: Radiation: brachytherapy

INTERVENTIONS:
Radiation: brachytherapy — An experimental arm using MRI imaging and excluding the transition zone from the target volume
  Groups: MRBT
Radiation: brachytherapy — Standard ultrasound-guided brachytherapy with standard target volumes
  Groups: USBT1
Radiation: brachytherapy — Standard ultrasound-guided brachytherapy with standard target volumes
  Groups: USBT2

SUMMARY:
The purpose of this research study is to assess outcomes of treatment for early prostate cancer. Current treatments for early (non-metastatic) cancer may cause long-term impairments in the patients quality of life. In this study we will compare the outcomes of patients treated with two alternative brachytherapy (seed implants) techniques using a series of questionnaires.

DETAILED DESCRIPTION:
Participants will be asked to complete a questionnaire about their health prior to treatment, at 1, 3 and 12 months after treatment and then once a year 4 more times.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of an adenocarcinoma of the prostate
* 18 years of age or older
* Prior choice of either standard brachytherapy or MRIGPB as primary treatment

Exclusion Criteria:

* Prior primary therapy (surgery or external beam radiation) for prostate cancer
* Current hormone ablation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have indicated their intention to receive brachytherapy at one of the four accrual sites.
Sampling Method: Non-Probability Sample
Enrollment: 414 (Estimated)
Dates: Start 2002-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
To assess changes in generic and disease specific quality of life over time after treatment with brachytherapy for early prostate cancer | 10 years

SECONDARY OUTCOMES:
To compare these outcomes after two alternative brachytherapy techniques, standard ultrasound guided brachytherapy and MRI guided prostate brachytherapy (MRIGPB) | 10 years
To identify factors associated with specific adverse outcomes. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: James Talcott, MD, SM, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute/Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts